CLINICAL TRIAL: NCT03944863
Title: Impact of Antibiotic Prophylaxis and Conditioning Modalities in Per Oral Endoscopic Myotomy for Esophageal Motor Disorders
Brief Title: Impact of Antibiotic Prophylaxis in Per-oral Endoscopic Myotomy for Esophageal Motor Disorders
Status: Completed | Type: Observational
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, VANBIERVLIET, Medical Doctor,Physician Doctor, Principal Investigator, Société Française d'Endoscopie Digestive
Other Study IDs: Antibiotic Prophylaxis POEM
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Esophagus Disorder; Esophageal Achalasia
Keywords: antibiotic prophylaxis; per oral endoscopic myotomy
MeSH Terms: conditions — Esophageal Diseases; Esophageal Achalasia | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- POEM + Antibiotic prophylaxis: Cefazolin: 2g or Amoxicillin - clavulanic acid: 1g x 3 during 7 days
  Interventions: Drug: Antibiotics
- POEM + No antibiotic prophylaxis

INTERVENTIONS:
Drug: Antibiotics
  Groups: POEM + Antibiotic prophylaxis

SUMMARY:
No recommendation regarding antibiotic prophylaxis and preparation modalities are available for patients with esophageal motor disorders who benefit from Per-Oral Endoscopic Myotomy (POEM). The aim of our study was to evaluate the impact of antibiotic prophylaxis on the POEM's safety.

This study was a comparative and multicentric retrospective analysis of a database prospectively maintained. Patients over 18 year's old with esophageal motor disorders confirmed by prior manometry, who underwent POEM were included. The primary endpoint was the occurrence of complications, as classified by Cotton, based on whether or not antibiotic prophylaxis was administered.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients presenting a major esophageal motor disorder confirmed by prior manometry according to the Chicago classification and treated by per-oral endoscopic myotomy after a multidisciplinary meeting decision

Exclusion Criteria:

* Under-age patients were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients presenting a major esophageal motor disorder confirmed by prior manometry according to the Chicago classification and treated by per-oral endoscopic myotomy after a multidisciplinary meeting decision. Under-age patients were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2013-12; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The occurence of postoperative complications, according to Cotton's classification | 7 Days
  Depending on whether or not antibiotic prophylaxis was administered

SECONDARY OUTCOMES:
The evaluation of the efficacy of the procedure | 1 Month
  According to the Eckard score
The occurence of perioperative and postoperative complications | 7 Days
  According to Cotton's classification
The C-Reactive Protein and white blood cells count sampled | 1 Day
  Blood test the day after the procedure, level of CRP in mg/L

IPD SHARING:
Plan to Share IPD: Undecided